CLINICAL TRIAL: NCT00199251
Title: A 6-Week Multicentre, Double-Blind, Randomised, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy and Safety of Rupatadine 10 and 20 Mg in the Treatment of Chronic Idiopathic Urticaria (CIU): a Phase III Clinical Trial
Brief Title: Efficacy and Safety of Rupatadine 10 and 20 Mg in Chronic Idiopathic Urticaria
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: J. Uriach and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IC010RUP304
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-12-23 (Estimated); Status verified 2005-09

CONDITIONS: Urticaria
Keywords: URTICARIA, WHEALS, FLARE, ANTIHISTAMINE, ANTIHISTAMINE
MeSH Terms: conditions — Urticaria | interventions — rupatadine

INTERVENTIONS:
Drug: RUPATADINE

SUMMARY:
· To evaluate the efficacy of rupatadine 10 and 20 mg for the treatment of CIU symptoms over four-week treatment period in comparison with placebo.

DETAILED DESCRIPTION:
STUDY PHASE III OBJECTIVES · To evaluate the efficacy and safety of rupatadine 10 mg and 20 mg for the treatment of CIU symptoms over four-week treatment period in comparison with placebo.

DESIGN · A multicentre, double blind, randomised, placebo controlled, parallel-group study in 300 patients (100 patients each treatment) group.

INDICATION · Chronic Idiopathic Urticaria (CIU) ASSESSMENT Primary efficacy measure of each treatment will compare the frequency and severity of symptoms of CIU as measured by the patient in terms of change in mean pruritus score (MPS) over the 4-week treatment period.Secondary efficacy measures include change from baseline over the 4 and 6-week treatment period in the mean number of wheals (MNW) score; mean total symptoms score (MTSS), calculated as the sum of the MPS (Mean pruritus symptoms) and the MNW (Mean number of wheals) scores, severity of symptoms of CIU as measured by the patient in terms of change in mean pruritus score (MPS) over the 6-week treatment period, Visual Analogic Scale (VAS) and Quality of life (QoL) which will be assessed by the "Dermatology Life Quality Index" (DLQI).Safety: ECGs baseline and final visit; clinical laboratory controls, physical examination, incidence of adverse events (AE).

STUDY POPULATION 300 patients between 12-65 years of age, with CIU

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman aged between 12 and 65
2. Active CIU (score ³2 labeled as moderate pruritus) for at least 3 days (not necessarily consecutive days) in the week before inclusion with a total score of active CIU ³6 labeled as moderate pruritus for these 3 days
3. Documented history of active CIU (urticaria wheals) with or without an associated angioedema for at least three days per week over the last 6 weeks prior to Screening Visit.
4. 12 lead ECG obtained at screening within acceptable limits, moreover in absence of any drug effect or disease, QTc interval values (msec) after Bazzet's correction must be normal (not prolonged). The values considered to be normal are < 430 msec for males and < 450 msec for females.
5. Patient who signed the informed consent form. In case the patient to be underage (from 12 to 18, -and 21 for Argentina-) the written informed consent of one of his/her parents or legal guardian is required.
6. Women of childbearing potential should have a negative pregnancy test at the time of inclusion. In addition, they must use an effective contraceptive method (i.e. oral, IUD, condom, etc). The commitment of the patient to use these measures while participating in this clinical trial will be considered as sufficient.

Exclusion Criteria:

1. CIU associated to some underlying disease (Hodgkin's disease/vasculitis/lupus erythematous/hepatitis)
2. Patient under any systemic or topical medication for CIU and/or an inferior wash-out period as stated as follows:

   * H1-receptor antagonists: fexofenadine (5 days prior to Day 0), loratadine, desloratadine, cetirizine, hydroxyzine, diphenhydramine, cyproheptadine, etc. (3 days prior to Day 0)
   * H2-receptor antagonists: cimetidine, ranitidine, famotidine, etc (2 days prior to Day 0)
   * H1- and H2-receptor antagonists: doxepin (7 days prior to Day 0)
   * Leukotriene antagonists: zafirlukast, montelukast, etc (4 days prior to Day 0)
   * Corticosteroids: prednisone, methylprednisolone, etc ( 28 days prior to Day 0)
   * Tricyclic antidepressants: imipramin, amitriptilin, etc (30 days prior to Day 0)

   The informed consent form must be signed prior to any washout period is set up.
3. Patients with analytical values twice as high than the upper limit of normality in the following parameters: ALP, ALT, AST, GGT and creatinine, and 1,5 times higher for than the upper limit of normality for the CK. Any other laboratory relevant finding should be assessed by the investigator before patient inclusion.
4. Cholinergic urticaria.
5. Patient taking medication that is known to interact with CYP3A4 isozyme of cytochrome P450 such as amiodarone, carbamazepine, cyclosporin, terfenadine, glucocorticoids, phenytoin, rifampicin, macrolides (e.g. erythromycin,clarytomicine, etc) and antifungal (e.g. ketoconazole, miconazole, fluconazole, etc) as well as grapefruit juice.
6. Urticaria due to known etiology (e.g. medications, insects bites, food, cold/heat, sun, etc)
7. Patient that after review of his medical history, is considered by the investigator as unresponsive to antihistaminic treatment
8. Pregnant or lactating female
9. Patients who are currently participating in or have participated in another clinical trial within the last three months
10. Patients who have a recent history (within previous 12 months) of drug addiction or alcohol abuse
11. Patient taking drugs strongly associated with torsade de pointes such as disopyramide, procainamide, quinidine, amiodarone, sotalol, thioridazine, beperidil or prenylamine.
12. Patient under any other treatment that could lead to symptomatic relief of the urticaria symptoms, for example: creams, lotions, ointments, homeopathy, etc… with or without recognized active ingredient.

(../.)

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2004-04; Study Completion 2005-06

PRIMARY OUTCOMES:
· To evaluate the efficacy of rupatadine 10 and 20 mg for the treatment of CIU symptoms over four-week treatment period in comparison with placebo.

SECONDARY OUTCOMES:
· To evaluate the efficacy and safety of rupatadine 10 and 20 mg for the treatment of CIU symptoms over six-week treatment period in comparison with placebo.
· To evaluate the safety of rupatadine 10 and 20 mg for the treatment of CIU symptoms over four-week treatment period in comparison with placebo.
· To assess the patient discomfort by using a VAS.
· To assess the patient QoL by a specific questionnaire, the DLQI.

CONTACTS AND LOCATIONS:
Overall Officials: EVA ARNAIZ, PhD, Study Director — J. Uriach y Compañía